CLINICAL TRIAL: NCT00472992
Title: TYSABRI® Pregnancy Exposure Registry
Brief Title: Pregnancy Exposure Registry for Tysabri®
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS401
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Crohn's Disease; Prenatal Exposure; Multiple Sclerosis; Pregnancy
Keywords: Pregnancy; TYSABRI
MeSH Terms: conditions — Crohn Disease; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the Registry was to evaluate the outcomes of pregnancy in women with Multiple Sclerosis (MS) or Crohn's Disease (CD) who were exposed to TYSABRI® at any time within 90 days prior to first day of Last Menstrual Period (LMP) or during pregnancy.

DETAILED DESCRIPTION:
This study was conducted in coordination with the TYSABRI® Global Observational Program in Safety (TYGRIS) observational study in the United States (US), Canada, and Rest of World (ROW).

The Coordinating Center (CC) monitored participants throughout their pregnancies and monitored the infants until 8 to 12 weeks of age in the US and Canada, and within 4 weeks after the Estimated Date of Delivery (EDD) in the ROW.

ELIGIBILITY:
Key Inclusion Criteria:

Females who become pregnant while they are taking TYSABRI® as part of the TYGRIS program, during a clinical trial with TYSABRI® that is sponsored by Biogen-Idec, or in the post-marketing setting may enroll in this Registry, as follows:

1. Documentation that the patient was exposed to TYSABRI® within 90 days prior to first day of Last Menstrual Period (LMP) or during pregnancy. (If exposure dates are unknown, the reporter must be able to specify or estimate trimester of exposure).
2. The outcome of the pregnancy must not be known at the time of enrollment. For pregnancies for which the outcomes are known at the time of enrollment, the information will be collected as retrospective reports and analyzed separately.
3. For US patients, verbal informed consent must be collected at the time of enrollment. The Coordinating Center (CC) obtains verbal informed consent (if verbal consent has not already been obtained by the physician). The CC then mails the patient a Release of Medical Information form to sign and return. If the patient is a minor, verbal consent must be obtained from the parent or legal guardian and verbal assent must be obtained from the patient.
4. For Canadian patients, a written informed consent must be collected by the TYGRIS investigator at the time of enrollment. A Release of Medical Information form will also be signed by the patient and returned to the CC.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with MS or CD who were exposed to Tysabri® in the US, Canada, and the Rest of World within 90 days prior to their last menstrual period.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2007-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of spontaneous abortions, fetal losses including stillbirths, and ectopic pregnancies | Approximately 9 months
Number of elective or therapeutic pregnancy terminations | Approximately 9 months
Number of Live Births | 4 weeks after the estimated date of delivery
Number of Live Births with Birth Defects | 8-12 weeks post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- United BioSource Corporation, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Friend S, Richman S, Bloomgren G, Cristiano LM, Wenten M. Evaluation of pregnancy outcomes from the Tysabri(R) (natalizumab) pregnancy exposure registry: a global, observational, follow-up study. BMC Neurol. 2016 Aug 24;16(1):150. doi: 10.1186/s12883-016-0674-4. PMID 27552976